CLINICAL TRIAL: NCT02326142
Title: A Phase 2, Double-blind, Parallel Group, Randomised, Placebo Controlled, Proof of Concept Study to Assess the Safety and Efficacy of OBE001 After Oral Administration in Pregnant Women With Threatened Preterm Labour.
Brief Title: A Phase 2 Study of OBE001 Versus Placebo in the Delay of Preterm Birth
Acronym: TERM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrolment difficulties.
Sponsor: ObsEva SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-OBE001-016
Record Dates: First submitted 2014-12-22; First posted 2014-12-25 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Preterm Labor
Keywords: Premature Obstetric Labor; Premature Birth
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth | interventions — OBE001

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OBE001 (Experimental)
  Interventions: Drug: OBE001
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OBE001 — OBE001 dispersible tablets for a single oral dose a day for up to 7 days.
  Arms: OBE001
Drug: Placebo — Placebo dispersible tablets for a single oral dose a day for up to 7 days.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the efficacy of a single dose of OBE001, an oral oxytocin antagonist, given for up to 7 days to delay preterm birth by 7 days compared to placebo.

DETAILED DESCRIPTION:
The study will be a multi-centre, randomised, parallel group, double-blind, placebo-controlled study in pregnant women with threatened preterm labour between 34^0/7 and 35^6/7 weeks of gestation.

The study will be in 2 parts as follows:

* from screening until the day of delivery (including a treatment period up to seven days)
* a maternal and neonatal follow-up period from the day of delivery until 28 days post expected term date (or until 28 days post-delivery should this be later).

In addition, there will be an observational, safety follow-up of the infants for 2 years to evaluate developmental outcome.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age (GA) between 34^0/7 and 35^6/7 weeks.
* Subjects with symptoms of preterm labour.
* Subjects with a singleton pregnancy.

Exclusion Criteria:

* Foetal death in utero in current pregnancy or in previous pregnancy after gestational week 24 or expected high risk of foetal death in the current pregnancy.
* Any contraindications for the mother or the foetus to stop labour or prolong pregnancy or any maternal or foetal conditions likely to indicate iatrogenic delivery.
* Use of cervical cerclage or a pessary in situ in the current pregnancy.
* The Subject has any condition which in the opinion of the PI constitutes a risk or a contraindication for the participation of the subject in the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2016-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
EFFICACY ENDPOINTS: Incidence of women delivering within 7 days post first dose | within 7 days of first dose

SECONDARY OUTCOMES:
EFFICACY ENDPOINTS: Incidence of women delivering within 48 hours post first dose | within 48 hours of first dose
EFFICACY ENDPOINTS: Incidence of women delivering before gestational age 37^0/7 weeks | up to 3 weeks post first dose
EFFICACY ENDPOINTS: Progression of uterine contractions from pre-dose to 6 hours and 24 hours post first dose | up to 24 hours post first dose
  Contractions measured by tocodynamometry.
EFFICACY ENDPOINTS: Assessment of maternal and foetal exposure to OBE001 (Maternal plasma concentrations of OBE001) | up to 7 weeks post first dose
  Maternal plasma concentrations of OBE001 on Day 1 (2 hours post first dose), on Day 2 (pre-dose and 2 hours post-dose) on Day 3 (pre-dose), Day 7 (post-dose) and at the time of delivery. Umbilical cord plasma concentration of OBE001 at the time of delivery.

OTHER OUTCOMES:
SAFETY ENDPOINTS: Evaluation of the maternal safety of OBE001 (Maternal incidence of adverse events (AEs), treatment-emergent adverse events (TEAEs), clinically significant changes in laboratory safety tests, 12-lead ECGs morphology or vital signs) | up to 28 days post expected term date
  Maternal incidence of adverse events (AEs), treatment-emergent adverse events (TEAEs), clinically significant changes in laboratory safety tests, 12-lead ECGs morphology or vital signs from Day 1 until 28 days after birth or term whichever is later.
SAFETY ENDPOINTS: Evaluation of the foetal safety of OBE001 (clinically significant changes in growth retardation and/or foetal heart rate monitoring and/or Amniotic Fluid Indices (AFI) | up to 14 days post first dose or birth whichever is earlier
  Incidence of foetal distress as determined by clinically significant changes in growth retardation and/or foetal heart rate monitoring and/or Amniotic Fluid Indices (AFI) from Day 1 to Day 14 or birth, whichever is earlier
SAFETY ENDPOINTS: Evaluation of the newborn neonatal morbidity | up to 28 days post expected term date
  Incidence of infants experiencing adverse events assessed by vital signs, temperature, APGAR score, weight and head circumference at birth as well as measures of neonatal morbidity from birth until 28 days after birth or term whichever is later
SAFETY ENDPOINTS: Evaluation of infant neurodevelopmental outocme. | up to 2 years after birth
  Incidence of infants with one or more Ages and Stages Questionnaire-3 domain score(s) below the cutoff at 6, 12, and 24 months, adjusted for gestational age.

CONTACTS AND LOCATIONS:
Locations (23):
- Belgium (3):
  - Brussels
  - Leuven
  - Liège
- Germany (4):
  - Bayreuth
  - Düsseldorf
  - Tübingen
  - Ulm
- Poland (5):
  - Bialystok
  - Chorzów
  - Lodz
  - Ruda Śląska
  - Warsaw
- Spain (5):
  - Barcelona
  - El Palmar
  - Madrid
  - Vitoria-Gasteiz
  - Zaragoza
- Switzerland (4):
  - Basel
  - Bern
  - Geneva
  - Lausanne
- United Kingdom (2):
  - Leeds
  - London